CLINICAL TRIAL: NCT04744623
Title: Clinical Evaluation of New Treatment Strategy of Mucous Membrane Pemphigoid Using Large Dose of Prednisolone Plus Intra-lesional of Triamcinolone Acetonide Followed by Combination of Mycophenolate Mofetil, Dapsone and Low Dose Prednisolone
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, rehab ghouraba, lecturer, Tanta University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Benign Mucous Membrane Pemphigoid
MeSH Terms: conditions — Pemphigoid, Benign Mucous Membrane | interventions — Dapsone; Prednisolone

STUDY DESIGN:
Intervention Model Description: 10 patients suffering from MMP were selected after complete diagnosis based on their clinical diagnosis and immunopathologic findings of IgG, IgA, and/or C3 targeting skin basement membranes with a linear deposition pattern referred from dermatology department. These patient were treated using large dose of prednisone 60mg daily plus intrational injection of Triamcinolone Acetonide every week until no further improvement of the lesion occurred (stage I) then the prednisolone is withdrawn gradually and substituted with using 1 g of MMF plus 50 mg dapsone till the lowest dose of prednisone could be reached (stage II). The lesion size and pain score will be assessed before treatment and during treatment in stage I and stage II. These data will be tabulated and statistically analyzed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- effect of large dose corticosteroids with intra-lestional injection in treatment of MMP (Experimental): 10 patients suffering from MMP were selected referred from dermatology department. These patient were treated using large dose of prednisone 60mg daily plus intra-lesion injection of Triamcinolone Acetonide every week until no further improvement of the lesion occurred (stage I)
  Interventions: Drug: large dose of prednisolone plus intra-lesional of Triamcinolone Acetonide followed the systemic combination of mycophenolate mofetil (MMF), dapsone and low dose prednisolone in treatment of MMP
- effect of of (MMF), dapsone and cortisone in treatment of MMP (Experimental): 10 patients suffering from MMP were selected referred from dermatology department. These patient were treated using large dose of prednisone 60mg daily plus intra-lesion injection of Triamcinolone Acetonide every week until no further improvement of the lesion occurred (stage I) then the prednisolone is withdrawn gradually and substituted with using 1 g of MMF plus 50 mg dapsone till the lowest dose of prednisone could be reached (stage II).
  Interventions: Drug: large dose of prednisolone plus intra-lesional of Triamcinolone Acetonide followed the systemic combination of mycophenolate mofetil (MMF), dapsone and low dose prednisolone in treatment of MMP

INTERVENTIONS:
Drug: large dose of prednisolone plus intra-lesional of Triamcinolone Acetonide followed the systemic combination of mycophenolate mofetil (MMF), dapsone and low dose prednisolone in treatment of MMP — 10 patients suffering from MMP were selected after complete diagnosis based on their clinical diagnosis and immunopathologic findings of IgG, IgA, and/or C3 targeting skin basement membranes with a linear deposition pattern refered from dermatology department. These patient were treated using large dose of prednisone 60mg daily plus intrational injection of Triamcinolone Acetonide every week until no further improvement of the lesion occurred (stage I) then the prednisolone is withdrawn gradually and substituted with using 1 g of MMF plus 50 mg dapsone till the lowest dose of prednisone could be reached (stage II).

SUMMARY:
Abstract: Mucous membrane pemphigoid (MMP) is an autoimmune blistering disorder characterized by inflammation, blistering, and scarring and predominantly occurring at mucous membranes. Successful treatment can be challenging, and uncontrolled disease may result in significant morbidity with scarring of the conjunctiva and oropharynx leading to blindness and dysphagia. Therefore successful treatment is a must to improve patient quality of life.

Aim of work: to evaluate clinically the effectiveness of systemic large dose of prednisolone plus intra-lesional of Triamcinolone Acetonide followed the systemic combination of mycophenolate mofetil (MMF), dapsone and low dose prednisolone in treatment of MMP cases.

Materials and method: 10 patients suffering from MMP were selected after complete diagnosis based on their clinical diagnosis and immunopathologic findings of IgG, IgA, and/or C3 targeting skin basement membranes with a linear deposition pattern refered from dermatology department. These patient were treated using large dose of prednisone 60mg daily plus intrational injection of Triamcinolone Acetonide every week until no further improvement of the lesion occurred (stage I) then the prednisolone is withdrawn gradually and substituted with using 1 g of MMF plus 50 mg dapsone till the lowest dose of prednisone could be reached (stage II). The lesion size and pain score will be assessed before treatment and during treatment in stage I and stage II. These data will be tabulated and statistically analyzed

DETAILED DESCRIPTION:
Before starting any treatment the size of the lesion will be measured and pain score will be evaluated. then patient were treated using large dose of prednisone 60mg daily plus intra-lesional injection of Triamcinolone Acetonide every week until no further improvement of the lesion occurred (stage I) at this stage the patients pain would be evaluated and lesion size would be measured .

as no further improvement is gained, the prednisolone is withdrawn gradually and substituted with using 1 g of MMF plus 50 mg dapsone till the lowest dose of prednisone could be reached (stage II) at this stage the patients pain would be evaluated and lesion size would be measured. then the data will be tabulated and statistically analyzed regarding pain score and lesion size

ELIGIBILITY:
Inclusion Criteria:

patients with age references patients confirmed from dermatology department that they had mucous membrane(MMP) pemphigoid- patients are not allergic o to the drugs being used for the treatment

Exclusion Criteria:

patients below or above age reference used in the study patients with other oral lesions not being confirmed as MMP patients with systemic diseases preventing using of the drugs

-

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-11-04 (Estimated)

PRIMARY OUTCOMES:
Mycophenolate mofetil, dapsone and low dose prednisolone may showing powerful effect than large dose of systemic corticosteroids with intra-lestional corticosteroid in treatment of Mucous membrane pemphigoid | from 10-11 months
  10 patients suffering from MMP were selected after complete diagnosis based on their clinical diagnosis and immunopathologic findings of IgG, IgA, and/or C3 targeting skin basement membranes with a linear deposition pattern refered from dermatology department. These patient were treated using large dose of prednisone 60mg daily plus intrational injection of Triamcinolone Acetonide every week until no further improvement of the lesion occurred (stage I) then the prednisolone is withdrawn gradually and substituted with using 1 g of MMF plus 50 mg dapsone till the lowest dose of prednisone could be reached (stage II).

SECONDARY OUTCOMES:
No difference in the effectiveness between large dose of prednisone with intra-lesional versus Mycophenolate mofetil, dapsone and low dose prednisolone | from 10-11 months
  10 patients suffering from MMP were selected after complete diagnosis based on their clinical diagnosis and immunopathologic findings of IgG, IgA, and/or C3 targeting skin basement membranes with a linear deposition pattern refered from dermatology department. These patient were treated using large dose of prednisone 60mg daily plus intrational injection of Triamcinolone Acetonide every week until no further improvement of the lesion occurred (stage I) then the prednisolone is withdrawn gradually and substituted with using 1 g of MMF plus 50 mg dapsone till the lowest dose of prednisone could be reached (stage II).

CONTACTS AND LOCATIONS:
Overall Officials: rehab f ghouraba, PHD, Principal Investigator — Tanta university, faculty of dentistry, Oral medicine clinic
Locations (1):
- Rehab Fouad Ghouraba, Tanta, Grabia, Egypt

IPD SHARING:
Plan to Share IPD: No